CLINICAL TRIAL: NCT02032472
Title: Efficiency Program Monitoring and Control of Hypertension Through Pharmacy Offices. APOF Project
Brief Title: Efficiency of Monitoring and Control Program of Hypertension Through Pharmacy Offices. APOF Project
Acronym: APOF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Institut Catala de Salut (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: APOF_IDIAP
Record Dates: First submitted 2013-12-23; First posted 2014-01-10 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Hypertension
Keywords: Blood Pressure Monitoring, Ambulatory; Arterial Pressure; Hypertension Controlled; Pharmacies
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Health Center (usual practice) (No Intervention): Controlling arterial pressure in the health center (a common practice is carried out)
- Collaboration of pharmacies (Experimental): Pharmacies cooperate in Measurement of Arterial Pressure of patients
  Interventions: Other: Measurement of Arterial Pressure

INTERVENTIONS:
Other: Measurement of Arterial Pressure — Pharmacies cooperate in measuring blood pressure of patients
  Arms: Collaboration of pharmacies

SUMMARY:
Background: Hypertension in adults is the factor most prevalent cardiovascular risk and motivates further inquiries, generating a very high cost of medical care.

Objective: To evaluate the monitoring of well-controlled hypertensive patients Pharmacy Offices. Hypothesis: the monitoring of these patients through the Office of Pharmacy will be as effective in obtaining good control of blood pressure as it is to obtained through health centers. Design: Multicenter randomized controlled trial along one year of follow up. Location: the city of Cerdanyola del Vallès (Barcelona). Participants: All patients diagnosed with hypertension and good control criteria in the past year. Arms: Health centers (control) and Pharmacy Offices (intervention). Outcome variable: blood pressure under good control along the monitoring

ELIGIBILITY:
Inclusion Criteria:

* Age not less than 18 years
* HTA controlled over 2 years of evolution
* Subjects with a history open to participating health centers or stable residence in the geographic area
* Subjects who agree to participate

Exclusion Criteria:

* Comorbidity and concomitant (Diabetes Mellitus, Heart failure or renal failure
* Patients with temporary residence in the geographic area of study
* Subjects of hypertension controlled by outside professionals to our primary care teams.
* Subjects with home care or any other cause which does not permit their displacement, transfer to the clinic or pharmacy during the evaluation period.
* Subjects with severe diseases of poor prognosis, hopefully less than one year of life.
* Subjects who do not have telephones.
* Subjects with communication problems (cognitive impairment, sensory, language barrier)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 677 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Percentage of hypertensive patients with criteria for good control of their arterial pressure along one year follow up | Monitoring of patients for 12 months (from January 1 to December 31, 2010)
  We considered as a for good control criterion , obtaining values of systolic arterial pressure to below 140 mm Hg and diastolic blood pressure below 90 mm Hg dea, held along the entire the year follow-up of patients

SECONDARY OUTCOMES:
reduction in the number of visits to the health center to measure blood pressure | Monitoring of patients for 12 months (from January 1 to December 31, 2010)
  The number of visits to the health center where blood pressure is measured. We hope that the number of visits to the health center where blood pressure is measured is lower in the intervention group (the patients have the option to go to the pharmacy to carrying out checks blood pressure)

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Solans, G Physician, Principal Investigator — Institut Català de la Salut (Spain)
Locations (1):
- Institut Català de la Salut (ICS), Cerdanyola Del Valllés, Barcelona, Spain